CLINICAL TRIAL: NCT03510845
Title: Arthroscopic Primary Repair of the Anterior Cruciate Ligament (ACL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1559
Record Dates: First submitted 2018-02-02; First posted 2018-04-27 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2018-02

CONDITIONS: Rupture of Anterior Cruciate Ligament
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Repairable ACL tear (Experimental): Patients whose ACL found to be avulsed from its femoral insertion or has a proximal tear, and intra-operatively, found to have a good tissue quality, will undergo arthroscopic ACL primary repair using fiberwires and SwiveLock screw to anchor the ligament into its origin, in the femoral condyle.
  Interventions: Procedure: Arthroscopic ACL Primary Repair
- Irreparable ACL tear (Other): Patients whose ACL cannot be repaired, will undergo arthroscopic ACL reconstruction using hamstring tendons.
  Interventions: Procedure: Arthroscopic ACL Reconstruction

INTERVENTIONS:
Procedure: Arthroscopic ACL Primary Repair — All patients (in both groups) will undergo diagnostic knee arthroscopy at the start of the procedure; those in the experimental arm "repairable ACL tear", whose ACL found to be avulsed from its femoral insertion or has a proximal tear, and intra-operatively, found to have a good tissue quality, will undergo arthroscopic ACL primary repair using fiberwires and SwiveLock screw to anchor the ligament into its origin, in the femoral condyle.
  Other Names: Diagnostic knee arthroscopy
  Arms: Repairable ACL tear
Procedure: Arthroscopic ACL Reconstruction — Patients whose ACL cannot be repaired, will undergo arthroscopic ACL reconstruction using hamstring tendons.
  Other Names: Diagnostic knee arthroscopy
  Arms: Irreparable ACL tear

SUMMARY:
A prospective cohort study that will be conducted at Sultan Qaboos University Hospital. It aims to determine the outcomes, in terms of, activity level, functional level, subjective knee function, range of motion, stability, and failure, among patients with acute ACL injuries, who undergo arthroscopic primary ACL repair; and to compare these results with patients who undergo arthroscopic ACL reconstruction. To the investigators' knowledge, there is a dearth of studies looking into the outcomes of arthroscopic primary ACL repair and this going to be the first study in the Middle East. The investigators believe that arthroscopic primary ACL repair is superior to arthroscopic ACL reconstruction; and conducting this research project will elucidate the previously abandoned facts about acute ACL repair; and will eventually have a huge impact in the field of orthopedic surgery.

DETAILED DESCRIPTION:
Hypothesis Null hypothesis: no difference in outcomes between arthroscopic primary ACL repair and arthroscopic ACL reconstruction in patients with acute ACL tear.

Alternative hypothesis: the arthroscopic primary ACL repair is superior to arthroscopic ACL reconstruction.

Background Anterior cruciate ligament (ACL) is an important mechanical stabilizer during knee-joint movement; it is the primary restraint against anterior tibial translation relative to the femur; and it acts as secondary restraint to tibial rotation and varus/valgus rotation. ACL injuries are commonly seen among athletics; and the number is increasing, with a reported incidence of 38/100,000 per year. Although there is still some debate about the optimal treatment for acute ACL tears, surgical management in the young and active patient is recommended. The surgical management options to an isolated ACL tear vary from acute repair to ligament reconstruction. Acute ACL repair can be classified into: acute primary repair, acute repair with the use of a ligament augmentation device, and acute repair with augmentation with an autologous hamstring tendon graft. The outcome of acute repair of ACL rupture from its femoral attachment or a proximal tear close to it, is the aim to be accomplished at the end of this project.

Several studies demonstrated that the results of acute repair of ACL ruptures deteriorate with time and the procedure was shown to be ineffective. However, most of the published studies are retrospective and nonrandomized, and they compare different surgical techniques, rehabilitation, and follow-up protocols. The surgeries were open and lengthy, the repairs were done on all injury types, on wide variety of ages, with varied concomitant injuries, and the rehab was primeval. Furthermore, there is no study that has described the long-term results of acute ACL repair.

Although the concept of ACL potential healing has been deserted in the past, there is renewed interest in the primary healing capacity of this ligament. One would argue why there is a need for the repair of a torn ACL. First, the operation is simple and takes less time and less risk in comparison to ACL reconstruction. Second, ACL treatment aims to provide immediate knee stability; resolve the pain and avoiding long-term complications, primarily osteoarthritis. ACL reconstruction using an autologous or allogenic tendon graft, is universally accepted as the gold standard treatment for complete ACL tears, as it yields excellent results for instability and pain in most the patients. However, there is a higher failure rate in adolescents than in other age groups with up to 20% to 25% of patients experiencing problems postoperatively. This mandates to find a better solution for this group of patients. In addition, patients post ACL reconstructions were found to have higher rates of osteoarthritis, despite the treatment; these findings are based on long-term follow up studies. This emphasizes on the need to find an alternative surgical management option to improve the ultimate outcomes. Third, the incidence of ACL injuries in skeletally immature patients are increasing; and so far, there are no standardized treatment options. For this group of patients, the transphyseal ACL reconstruction with grafts carries a risk for limb length and angular deformities, although several studies have proven no increase in the rate of such complications. Hence, the pre-pubescent population has the potential to benefit greatly from this regenerative treatment, which does not violate the physes; and they respond remarkably to certain biological stimuli implemented in the current enhanced repair techniques. Fourth, regeneration of the ACL over reconstruction preserves the remaining proprioceptive fibers within the ligament substance, and maintains the complex insertion sites of the ligament. This could potentially lead to more normal biomechanics of the knee if adequate regeneration is achieved.

Material and methods This is a prospective cohort study that will be conducted at Sultan Qaboos University Hospital (SQUH) and it involves patients with acute ACL injury attending the orthopedic clinic. The ACL rupture will be assessed clinically by anterior drawer test (ADT), Lachman's test, and pivot shift test. The ACL tear will be confirmed by knee MRI.

The ethical approval and permission from the concerned institution is required to start the study. All eligible patients who consent to participate will be included in the study.

The arthroscopic ACL repair will be carried out by one expert orthopedic surgeon. Because arthroscopy is a reference standard for the diagnosis of internal derangements of the knee, and because it is unethical to sacrifice a torn ACL that can be repaired; the patients will be assessed intra-operatively, and will be divided into two groups (group 1= ACL repair); group 2= ACL reconstruction) based on ACL amenability for repair or reconstruction. If the ACL was found to have a good tissue quality and fulfilling the inclusion criteria, it will be repaired using fiberwires and anchored to the femoral condyle using SwiveLock screw. If the ACL found irreparable, then it will be reconstructed using hamsting tendons graft. A minimum of 20 patients will be included in each group.

Post-operatively, the patients will undergo a specific rehabilitation program and will be followed up for, at least, one year to determine their activity level, functional level, subjective knee function, range of motion, stability, and failure of the repair.

The activity level will be evaluated using Tegner activity score, which is a scale that aims to provide a standardized method of grading work and sporting activities. It describes the current level of activity and that before injury. The score varies from 0-10; a score of 0 represents sick leave or disability pension because of knee problems, whereas a score of 10 corresponds to participation in national and international elite competitive sports.

The functional state will be graded using Lysholm scale, which is designed to assess how the knee problems have affected the patient's ability to manage in everyday life. It consists of 8 items that assess: pain (25 points), instability (25 points), locking (15 points), swelling (10 points), limp (5 points), stair climbing (10 points), squatting (5 points), and need for support (5 points). Every question response has been assigned an arbitrary score on an increasing scale. The total score is the sum of each response to the eight questions, and may range from 0-100. The scores are categorized as: Poor (<65); Fair (65-83); Good (84-90); and Excellent (>90).

Both scales will be translated into Arabic; then back-translation will be done into English, all by experts, to ensure absolute quality and accuracy.

The subjective knee function will be graded as poor, fair, good, and excellent.

The knee stability/anterior laxity will be assessed using ADT, Lachman's test, and pivot shift test. The ADT is graded as:

* Negative (0)
* +1: <5 mm translation,
* +2: 5 to 10 mm,
* +3: >10 mm translation.

The Lachman's test is graded as:

* Negative (0),
* Slight (1+): <5 mm of displacement,
* Moderate (2+): 5 to 10 mm,
* Severe (3+): >10 mm compared with that of the normal knee.

The pivot shift is graded as:

* Negative (0)
* Trace positive (1+),
* Moderate shift (2+),
* Subluxation (3+).

The patients will be evaluated by an independent observer.

The participants' data, including the personal information, will be kept safe and secure. The date will be anonymised with ID numbers. The hard copies will be in a locked filing cabinet and the soft copies will be securely password protected. The data will only be accessed by the agreed members of the research team. These records are not to be transferred to or shared with any other institute.

The Statistical Package for the Social Sciences (SPSS) will be used for the statistical analyses. Data collection and entry will be done by trained personnel. To assess relationship between variables: as univariate analysis, we will use Chi-square, t-test, ANOVA or non-parametric tests according to the nature of data. The nonparametric analysis of variance (Kruskal-Wallis test) will be used to determine the significance of the overall difference in the outcome measures among the two groups at a particular follow-up time-point. Paired comparisons among the two groups at each time-point will be made with use of the Mann-Whitney test. The Wilcoxon test for paired data will also be used to test for the significance of the changes in the outcome measures for a particular group between any two time points. Also, odd ratio will be calculated, where applicable. As adjusted multivariate analysis, we will use logistic regression. Relations between variables will be assessed by correlation coefficient.

Feasibility of the project This study is going to be a pilot study. Its primary mission is to provide immediate knee stability, resolve the pain and avoid long-term complications via simple and straightforward arthroscopic ACL repair. It is an evolving procedure and its results are promising. ACL injuries are common and the procedures are being done by one experienced orthopedic surgeon. The assessment scales that will be used are validated and have been used internationally in previous studies yielding valid information. To the investigator's knowledge, there is a dearth of studies looking into the outcomes of arthroscopic primary ACL repair and this is going to be the first study in the Middle East. Therefore, conducting this research project will yield reliable and helpful results; will elucidate the previously abandoned facts about acute ACL repair; and will eventually have a huge impact in the field of orthopedic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Acute ACL injuries. i.e., within 3 month.
* ACL rupture from its femoral attachment or a proximal tear close to it
* Concomitant meniscal injuries

Exclusion Criteria:

* Chronic ACL injuries
* Mid-substance ACL tears
* Previous surgery on the injured knee
* Associated knee pathology (e.g. infection; fractures, osteoarthritis, etc).

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Activity level | 2 years
  Assessment of activity level by Tegner score. it describes preinjury & current activity level. The score varies from 0-10: 0 represents sick leave/disability pension because of knee problems while 10 corresponds to participation in national/international elite competitive sports.

SECONDARY OUTCOMES:
Functional level | 2 years
  Assessment of functional level by Lysholm score. It consists of 8 items assessing pain, instability, locking, swelling, limp, stair climbing, squatting & need for support. It ranges from 0-100 & is categorized as Poor <65; Fair 65-83; Good 84-90; & Excellent>90.

OTHER OUTCOMES:
Subjective knee function | 2 years
  It is patient reported & is graded as poor, fair, good, & excellent.
Knee stability | 2 years
  Assessed by stability tests, which are anterior drawer, Lachman & pivot shift tests. The ADT and Lachman are graded as -ve 0; +1: <5 mm translation, +2: 5-10 mm, +3: >10 mm. The pivot shift is graded as -ve 0; Trace +ve 1+, Moderate shift 2+ & Subluxation 3+.
Knee range of motion | 2 years
  Assessed by using a goniometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Sultan Qaboos University Hospital, Muscat, Oman

IPD SHARING:
Plan to Share IPD: No
A full manuscript write-up will be shared at the end of the study.

REFERENCES:
- [Background] Rupp S, Kaltenkirchen N, Hopf T, Gleitz M. [Clinical relevance of tunnel position and interference screw location after replacement-plasty of the anterior cruciate ligament with a patellar ligament transplant]. Unfallchirurg. 1995 Dec;98(12):650-4. German. PMID 8584948
- [Background] Feagin JA Jr, Curl WW. Isolated tear of the anterior cruciate ligament: 5-year follow-up study. Am J Sports Med. 1976 May-Jun;4(3):95-100. doi: 10.1177/036354657600400301. PMID 984289
- [Background] Andersson C, Gillquist J. Treatment of acute isolated and combined ruptures of the anterior cruciate ligament. A long-term follow-up study. Am J Sports Med. 1992 Jan-Feb;20(1):7-12. doi: 10.1177/036354659202000103. PMID 1554077
- [Background] Andersson C, Odensten M, Gillquist J. Knee function after surgical or nonsurgical treatment of acute rupture of the anterior cruciate ligament: a randomized study with a long-term follow-up period. Clin Orthop Relat Res. 1991 Mar;(264):255-63. PMID 1997243
- [Background] Gluckert K, Kladny B, Blank-Schal A, Hofmann G. MRI of the knee joint with a 3-D gradient echo sequence. Equivalent to diagnostic arthroscopy? Arch Orthop Trauma Surg. 1992;112(1):5-14. doi: 10.1007/BF00431036. PMID 1482622
- [Background] Engstrom B, Gornitzka J, Johansson C, Wredmark T. Knee function after anterior cruciate ligament ruptures treated conservatively. Int Orthop. 1993;17(4):208-13. doi: 10.1007/BF00194180. PMID 8407034
- [Background] Radford WJ, Amis AA, Heatley FW. Immediate strength after suture of a torn anterior cruciate ligament. J Bone Joint Surg Br. 1994 May;76(3):480-4. PMID 8175860
- [Background] Odensten M, Lysholm J, Gillquist J. Suture of fresh ruptures of the anterior cruciate ligament. A 5-year follow-up. Acta Orthop Scand. 1984 Jun;55(3):270-2. doi: 10.3109/17453678408992354. PMID 6377805
- [Background] Sommerlath K, Lysholm J, Gillquist J. The long-term course after treatment of acute anterior cruciate ligament ruptures. A 9 to 16 year followup. Am J Sports Med. 1991 Mar-Apr;19(2):156-62. doi: 10.1177/036354659101900211. PMID 2039067
- [Background] Fruensgaard S, Kroner K, Riis J. Suture of the torn anterior cruciate ligament. 5-year follow-up of 60 cases using an instrumental stability test. Acta Orthop Scand. 1992 Jun;63(3):323-5. doi: 10.3109/17453679209154792. PMID 1609600
- [Background] Mohtadi N, Grant J. Managing anterior cruciate ligament deficiency in the skeletally immature individual: a systematic review of the literature. Clin J Sport Med. 2006 Nov;16(6):457-64. doi: 10.1097/01.jsm.0000248844.39498.1f. PMID 17119358
- [Background] Daniel DM, Stone ML, Dobson BE, Fithian DC, Rossman DJ, Kaufman KR. Fate of the ACL-injured patient. A prospective outcome study. Am J Sports Med. 1994 Sep-Oct;22(5):632-44. doi: 10.1177/036354659402200511. PMID 7810787
- [Background] Lohmander LS, Roos H. Knee ligament injury, surgery and osteoarthrosis. Truth or consequences? Acta Orthop Scand. 1994 Dec;65(6):605-9. doi: 10.3109/17453679408994613. PMID 7839844
- [Background] von Porat A, Roos EM, Roos H. High prevalence of osteoarthritis 14 years after an anterior cruciate ligament tear in male soccer players: a study of radiographic and patient relevant outcomes. Ann Rheum Dis. 2004 Mar;63(3):269-73. doi: 10.1136/ard.2003.008136. PMID 14962961
- [Background] Lohmander LS, Englund PM, Dahl LL, Roos EM. The long-term consequence of anterior cruciate ligament and meniscus injuries: osteoarthritis. Am J Sports Med. 2007 Oct;35(10):1756-69. doi: 10.1177/0363546507307396. Epub 2007 Aug 29. PMID 17761605
- [Background] Wester W, Canale ST, Dutkowsky JP, Warner WC, Beaty JH. Prediction of angular deformity and leg-length discrepancy after anterior cruciate ligament reconstruction in skeletally immature patients. J Pediatr Orthop. 1994 Jul-Aug;14(4):516-21. doi: 10.1097/01241398-199407000-00019. PMID 8077439
- [Background] Koman JD, Sanders JO. Valgus deformity after reconstruction of the anterior cruciate ligament in a skeletally immature patient. A case report. J Bone Joint Surg Am. 1999 May;81(5):711-5. doi: 10.2106/00004623-199905000-00014. No abstract available. PMID 10360701
- [Background] Cohen DJ, Kim D, Baim DS. Origin of the left main coronary artery from the "non-coronary" sinus of Valsalva. Cathet Cardiovasc Diagn. 1991 Mar;22(3):190-2. doi: 10.1002/ccd.1810220308. PMID 2013083
- [Background] Henry J, Chotel F, Chouteau J, Fessy MH, Berard J, Moyen B. Rupture of the anterior cruciate ligament in children: early reconstruction with open physes or delayed reconstruction to skeletal maturity? Knee Surg Sports Traumatol Arthrosc. 2009 Jul;17(7):748-55. doi: 10.1007/s00167-009-0741-0. Epub 2009 Feb 28. PMID 19252897
- [Background] Trentacosta NE, Vitale MA, Ahmad CS. The effects of timing of pediatric knee ligament surgery on short-term academic performance in school-aged athletes. Am J Sports Med. 2009 Sep;37(9):1684-91. doi: 10.1177/0363546509332507. Epub 2009 May 21. PMID 19460815
- [Background] Mastrangelo AN, Haus BM, Vavken P, Palmer MP, Machan JT, Murray MM. Immature animals have higher cellular density in the healing anterior cruciate ligament than adolescent or adult animals. J Orthop Res. 2010 Aug;28(8):1100-6. doi: 10.1002/jor.21070. PMID 20127960
- [Background] Mastrangelo AN, Magarian EM, Palmer MP, Vavken P, Murray MM. The effect of skeletal maturity on the regenerative function of intrinsic ACL cells. J Orthop Res. 2010 May;28(5):644-51. doi: 10.1002/jor.21018. PMID 19890988
- [Background] Vavken P, Murray MM. Translational studies in anterior cruciate ligament repair. Tissue Eng Part B Rev. 2010 Feb;16(1):5-11. doi: 10.1089/ten.teb.2009.0147. PMID 20143926
- [Background] Drogset JO, Grontvedt T, Robak OR, Molster A, Viset AT, Engebretsen L. A sixteen-year follow-up of three operative techniques for the treatment of acute ruptures of the anterior cruciate ligament. J Bone Joint Surg Am. 2006 May;88(5):944-52. doi: 10.2106/JBJS.D.02876. PMID 16651567
- [Background] DiFelice GS, van der List JP. Arthroscopic Primary Repair of Proximal Anterior Cruciate Ligament Tears. Arthrosc Tech. 2016 Sep 19;5(5):e1057-e1061. doi: 10.1016/j.eats.2016.05.009. eCollection 2016 Oct. PMID 27909675